CLINICAL TRIAL: NCT00312637
Title: High-Resolution Axillary MRI With Magnetic Resonance Spectroscopy as a Non-Invasive Test for Determining Pathologic Lymph Node Status in Patients With Invasive Breast Cancer
Brief Title: Using Magnetic Resonance Spectroscopy With MRI to Non-invasively Determine Breast Cancer Extent of Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC0426
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Staging
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopy

SUMMARY:
The purpose of this study is to evaluate whether high-resolution magnetic resonance imaging of the axilla with spectroscopy can identify nodal features suggestive of metastatic involvement in patients diagnosed with invasive breast cancer. This may enable us to define a select group of patients for whom axillary lymph node dissection could be avoided.

DETAILED DESCRIPTION:
Breast cancer is the second leading cause of death in women. The spread of cancer from the breast to the lymph nodes is a significant factor in determining breast cancer survival. Currently, surgical procedures are performed to determine lymph node involvement. Full axillary lymph node dissection has a high morbidity associated with the procedure. While sentinel lymphadenectomy avoids a full axillary dissection in clinically negative axilla in untreated patients, it has been reported to have a false negative rate of less than 10%. Others have reported higher false negative rates after neoadjuvant chemotherapy. For those reasons, there is considerable interest in non-invasive methods that may allow staging of the axilla.

Magnetic resonance imaging (MRI) of the breast with contrast-enhancement is increasingly being used in breast cancer patients to determine the size of the tumor and its extent. A few reports from Europe have been published regarding its use in evaluating axillary lymph node metastases preoperatively, and the results appear promising. Kvistad et al. demonstrated lymph node metastases using dynamic contrast-enhanced MRI, in which the study had a sensitivity of 83%, a specificity of 90%, and an accuracy of 88%. Luciani et al, suggest that lymph nodes with a large size, irregular contours, round hila, high-signal intensity on T2 sequences, and those with marked enhancement are associated with malignancy.

Magnetic resonance imaging with spectroscopy (MRS) has been used in clinical practice for evaluation of brain tumors as a method for noninvasive detection of tumor metabolism. More recently, it has been used on other soft-tissue tumors, including breast. Like other soft-tissue tumors, breast cancers have increased levels of the amino acid choline. In several studies, the sensitivity and specificity of MRS for detecting breast cancer ranged from 73%-92% and 71%-93%, respectively. No known MRS data has been published regarding axillary lymph node involvement in patients with breast cancer. It is postulated that the choline peak should be elevated in lymph nodes with metastatic breast cancer.

This is an observational study. All eligible patients who give informed consent will complete a MRI/MRS screening questionnaire and if there are no contraindications will undergo MRI/MRS imaging prior to their clinically indicated sentinel lymphadenectomy which may be followed by axillary dissection to be determined by surgeon during the course of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with recent (within 60 days) invasive breast cancer.
* No previous ipsilateral axillary surgery.

Exclusion Criteria:

* Patients diagnosed with in situ disease.
* Patients with previous ipsilateral axillary surgery.
* Patients with MRI/MRA contraindications such as a cardiac pacemaker, an aneurysm clip, cochlear implants, and metal in the eyes.
* Patients who have had a moderate or severe contrast reaction to intravenous gadolinium-DTPA.
* Patients who are clinically not stable.
* Patients who cannot give consent.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherie M Kuzmiak, D.O., Principal Investigator — Department of Radiology, University of North Carolina at Chapel Hill
Locations (1):
- Mammography Clinic - UNC Hospitals, Chapel Hill, North Carolina, United States